CLINICAL TRIAL: NCT06024135
Title: Safety and Efficacy Assessments of NeoKidney®, a New Sorbent-based Hemodialysis Device, in ESRD Patients Treated With Short Daily Hemodialysis: a First in Human Use.
Brief Title: Safety and Efficacy Assessments of NeoKidney® in ESRD Patients Treated With Short Daily Hemodialysis
Acronym: FIH Caen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nextkidney S.A. (Industry)
Collaborators: Monitoring Force Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKH-CI22-01
Record Dates: First submitted 2023-08-16; First posted 2023-09-06 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-08

CONDITIONS: End Stage Renal Disease; ESRD
Keywords: Dialysis; Hemodialysis; Sorbent; Short daily hemodialysis; SDHD; HD; ESRD; End stage renal disease; Dialysate
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeoKidney therapy (Experimental): Every patient will receive NeoKidney therapy which will be referenced to SDHD sessions with the usual device as their own baseline.
  The study is designed in a way that allows an incremental increase of the ratio of NeoKidney versus SDHD sessions with the usual device. In order to minimize the study burden to the patient, most SDHD sessions with the usual device will be done in the patient's home. The NeoKidney therapy sessions, and 2 SDHD sessions with the usual device will be performed in the study center, thus ensuring the necessary patient care and observation as well as sample collection.
  Interventions: Device: NeoKidney

INTERVENTIONS:
Device: NeoKidney — Progressive exposition to NeoKidney device starting with only one NeoKidney therapy on a mid-week day and 5 SDHD sessions with the usual device in week one, followed by 2 NeoKidney therapies and 4 SDHD sessions with the usual device in week 2, and only progressing to a full week on NeoKidney after a safety review.

SUMMARY:
The goal of this clinical investigation is to asses the safety and efficacy a new sorbent-based hemodialysis device, NeoKidney® in ESRD patients treated with short daily hemodialysis.

Participants (stable SDHD patients) will undergo hemodialysis treatement on the NeoKidney® device at the hospital on a progressive exposition to the device:

* The first week, patient will be treated once with NeoKidney® on Wednesday
* The 2nd week the patient will be treated two consecutive days with NeoKidney® (in the middle of the week)
* On the 3rd week, after approval by the DSMB, the patients will be treated 6 consecutive days, in hospital, with the NeoKidney

All the other sessions will be performed with the patient's usual SDHD device at home except for two sessions prior to NeoKidney® sessions at Week 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or over;
2. Treated with short-daily hemodialysis (1.5-3 h sessions) 5-6 times a week for at least 3 months;
3. Estimated Urea removal concentration between [220 to 550] mmol. (Estimation based on the formula: ([Dry Weigh in kg]*] x 0,6)*([) x ([Last pre-dialysis urea concentration in mmol/L]*] x 0,5).
4. Well-functioning vascular access (native fistula or graft or permanent veinous catheter) defined as:

   * Capable of providing a blood flow rate of ≥200 mL/min, AND
   * Absence of vascular access revision for at least 3 months
5. For females of reproducible age, negative urinary pregnancy test and use of appropriate birth control method(s);
6. Ability to understand the informed consent and give informed consent;
7. Willingness and ability to comply with study procedures and to attend all study follow up visits

Exclusion Criteria:

1. Post-dialysis body weight below 41.0 kg
2. Hb <10.0 g/L, or pre-dialysis [Na] < 132 and > 145 mmol/L, pre-dialysis [K] < 3.5 and > 6 mmol/L and pre-dialysis [HCO3] < 15 and > 30 mmol/L in the latest determination, within the 6 weeks prior to enrollment.
3. One or more pre-dialysis urea concentration <10 mmol/L or >30mmol/L within the 6 weeks prior to enrollment.
4. Subjects requiring UF volume >2.0L per 2hr treatment in any dialysis session within 6 weeks prior to enrollment.
5. Any documented episode of hemolysis within the 6 months prior to enrolment.
6. Any infection related to the vascular access within the 4 weeks prior to enrolment.
7. History of impaired liver function (normal Factor V).
8. Severe uncontrolled arterial hypertension (systolic BP>180mmHg or diastolic BP >104 mmHg).
9. Known chronic obstructive pulmonary disease.
10. Anticipation of a living donor kidney transplantation within the 2 months of the study period.
11. Pregnant, breast feeding, or planning a pregnancy during the study period.

13. Any known psychosocial problems which may negatively influence dialysis treatment.

14. History of drug and/or alcohol abuse within the last 3 months prior to enrolment.

15. Patients with any serious medical condition which in the opinion of the investigator, may adversely affect the safety of the participant and/or effectiveness of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Absence of serious adverse events (SAE) and of serious adverse device effects (SADE). | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in patient's blood pressure (mm Hg) during treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on patient's clinical condition and vital parameters, in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in patient's heart rate (bpm) during treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on patient's clinical condition and vital parameters, in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in patient's body temperature (°C) during treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on patient's clinical condition and vital parameters, in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in patient's pulse oximetry (% SpO2) during treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on patient's clinical condition and vital parameters, in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in bicarbonates (mmol/L) pre- vs post-treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on hematology and clinical chemistry pre- vs post-treatment in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in pH pre- vs post-treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on hematology and clinical chemistry pre- vs post-treatment in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in LDH (UI/L) pre- vs post-treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on hematology and clinical chemistry pre- vs post-treatment in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in Haptoglobin (g/L) pre- vs post-treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on hematology and clinical chemistry pre- vs post-treatment in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in Sodium (mmol/L) pre- vs post-treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on hematology and clinical chemistry pre- vs post-treatment in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in Potassium (mmol/L) pre- vs post-treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on hematology and clinical chemistry pre- vs post-treatment in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in Phosphate (mmol/L) pre- vs post-treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on hematology and clinical chemistry pre- vs post-treatment in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in Calcium (mmol/L) pre- vs post-treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on hematology and clinical chemistry pre- vs post-treatment in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in Chlorine (mmol/L) pre- vs post-treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on hematology and clinical chemistry pre- vs post-treatment in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in Magnesium (mmol/L) pre- vs post-treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on hematology and clinical chemistry pre- vs post-treatment in a small number (n=3) of patients and HD sessions (9 sessions per patient).
Absence of critical change in Magnesium (µmol/L) pre- vs post-treatment | Through the end of last patient follow-up visit, an average of 2 months
  To assess the safety of the NeoKidney on hematology and clinical chemistry pre- vs post-treatment in a small number (n=3) of patients and HD sessions (9 sessions per patient).

CONTACTS AND LOCATIONS:
Overall Officials: Maxence Ficheux, Dr, Principal Investigator — University Hospital, Caen
Locations (1):
- CHU de Caen, Caen, Normandy, France